CLINICAL TRIAL: NCT01886794
Title: Role of Hormonal Status on Vascularization and Vaginal Tissue in Women With Pelvic Organ Prolapse
Brief Title: Hormonal Status on Blood Flow and Tissue in Pelvic Organ Prolapse
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Collaborator moved and not able to recreate full study team
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 13-114
Record Dates: First submitted 2013-06-14; First posted 2013-06-26 (Estimated); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Floor Disorders
Keywords: pelvic floor dysfunction; pelvic organ prolapse; vaginal estrogen effects
MeSH Terms: conditions — Pelvic Floor Disorders; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Postmenopausal, topical vaginal cream (Experimental): Postmenopausal participants randomized to topical vaginal cream containing estrogen or placebo for about one month's use prior to scheduled surgery. These will include those women randomized to estrogen cream.
  Interventions: Drug: Postmenopausal, topical vaginal estrogen cream
- Pre-menopausal, no topical vaginal cream (No Intervention): Pre-menopausal, no topical vaginal cream. These women will be examined at different stages in their menstrual cycle in order to compare characteristics of the cycle at high and lower estrogen timepoints.
- Postmenopausal, topical placebo cream (Placebo Comparator): Postmenopausal participants randomized to topical vaginal cream containing estrogen or placebo for about one month's use prior to scheduled surgery. These will include those women randomized to placebo.
  Interventions: Drug: Placebo Comparator: Postmenopausal, topical placebo cream

INTERVENTIONS:
Drug: Postmenopausal, topical vaginal estrogen cream — Topical vaginal estrogen cream is commonly but not universally used to improve the health of vaginal tissue prior to surgery. This study will provide data regarding estrogen effects for post-menopausal women undergoing pelvic organ prolapse.
  Other Names: Estrace vaginal cream
  Arms: Postmenopausal, topical vaginal cream
Drug: Placebo Comparator: Postmenopausal, topical placebo cream — Postmenopausal participants randomized to topical vaginal placebo for about one month's use prior to scheduled surgery.
  Other Names: Placebo vaginal cream
  Arms: Postmenopausal, topical placebo cream

SUMMARY:
Our primary aim in the current study is to determine important tissue differences, including muscle and connective tissue changes, between postmenopausal women and reproductive age women with pelvic floor dysfunction to help develop targeted and noninvasive treatments.

DETAILED DESCRIPTION:
Our primary aim in the current study is to determine important tissue differences, including muscle and connective tissue changes, between postmenopausal women and reproductive age women with pelvic floor dysfunction to help develop targeted and noninvasive treatments. We will perform in vivo evaluations with colposcopy and OCT to determine epithelial thickness and overall mucosal health prior to surgery. At the time of surgery, we will obtain tissue for histologic and imaging analysis.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 70 years of age
* Stage II or greater pelvic organ prolapse (POP)
* Individuals electing surgery to treat their POP
* Willing and able to comply with study procedures
* Willing and able to provide written informed consent

Exclusion Criteria:

* Contraindication for estrogen cream
* Any medical condition that in the opinion of the investigator would place the subject at increased risk for participation
* History of connective tissue disease
* Previous hysterectomy or pelvic organ prolapse surgery
* Known allergic reaction to any agent required by the protocol
* Use of hormone therapy in postmenopausal women in the last 90 days
* Pregnant or lactating females
* History of prior noncompliance or the presence or history of psychiatric condition that would in the opinion of the investigator make it difficult for the subject to comply with study procedures or follow instructions

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06-06 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Vincent, MD, Principal Investigator — UTMB Galveston
Locations (1):
- UTMB Galveston, Galveston, Texas, United States

REFERENCES:
- See also: Link to the clinic where recruitment will be performed — http://www.utmbhealth.com/PelvicHealth

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Postmenopausal, Topical Vaginal Cream | Pre-menopausal, no Topical Vaginal Cream | Postmenopausal, Topical Placebo Cream
Started | 2 | 3 | 2
Completed | 2 | 3 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postmenopausal, Topical Vaginal Cream | Pre-menopausal, no Topical Vaginal Cream | Postmenopausal, Topical Placebo Cream | Total
Number analyzed (Participants) | 2 | 3 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 1 | 5
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (4.5) | 44.7 (4.5) | 65.5 (1.5) | 56 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 3 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 2 | 2 | 2 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Epithelial Thickness
Description: Measure of vaginal epithelial thickness obtained by optical coherence tomography
Time Frame: Change in thickness visit 1 to visit 2 for the postmenopausal group (approximately 1 month apart), and change in thickness from follicular to luteal phase for premenopausal group (approximately 1 month apart).
Population: All participants who enrolled were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Postmenopausal, Topical Vaginal Cream | Pre-menopausal, no Topical Vaginal Cream | Postmenopausal, Topical Placebo Cream
Number analyzed (Participants) | 2 | 3 | 2
micrometers | 80 (23) | 25.5 (2.5) | -11 (5)

2. Secondary Outcome: Histologic Assessment of Excised Tissue
Description: Evaluated tissue samples obtained during surgery to examine collagen. Collagen score (Masson trichrome): 3=abundant collagen (dark blue stain), 2=collagen present (light blue stain), 1=scant collagen (minimal blue stain) Higher scores indicate more collagen, or better outcome. (note that study vaginal drug was stopped at visit 2 for postmenopausal subjects except in one subject who used active topical vaginal cream but stopped after 2 weeks due to AE. Her OCT score was obtained after 2 weeks of active cream, however the histology was obtained 2 weeks after discontinuation of study drug because Visit 2 was scheduled at the time of the AE and at the time of stopping the active cream. The OCT and histology results are not concordant due to being taken at different timepoints (visit 2 on active cream vs surgery 16 days later off cream)
Time Frame: 1 month after visit 1 (3-17days after visit 2)
Population: Histology was performed for the postmenopausal, topical vaginal cream, and the pre-menopausal, no topical vaginal cream group. There was no histology available from the 2 postmenopausal subjects randomly assigned to the placebo cream group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Postmenopausal, Topical Vaginal Cream | Pre-menopausal, no Topical Vaginal Cream | Postmenopausal, Topical Placebo Cream
Number analyzed (Participants) | 2 | 3 | 0
score on a scale | 2.0 (1.0) | 2.3 (0.5) |

ADVERSE EVENTS:
Time Frame: AE's were collected during the time the subjects were enrolled in the study, which was 4-6 weeks.
Arm/Group | Postmenopausal, Topical Vaginal Cream | Pre-menopausal, no Topical Vaginal Cream | Postmenopausal, Topical Placebo Cream
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 0/3 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Postmenopausal, Topical Vaginal Cream (N=2) | Pre-menopausal, no Topical Vaginal Cream (N=3) | Postmenopausal, Topical Placebo Cream (N=2)
Vulvovaginal discomfort/itching (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT01886794/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT01886794/ICF_001.pdf